CLINICAL TRIAL: NCT02517034
Title: Advancing Screening and Treatment for Older Patients With Cancer
Brief Title: Geriatric Assessment in Predicting Chemotherapy Toxicity and Vulnerabilities in Older Patients With Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15161; NCI-2015-01202 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15161 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-07-28; First posted 2015-08-06 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Solid Neoplasm
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (geriatric assessment-driven treatment) (Experimental): Patients follow an intervention plan created by the NP using the results of the geriatric assessment. The NP discusses the results of the assessment and treatment recommendations with the patient. They also share the treatment plan, proposed referrals, and specific vulnerabilities with the primary care physician and community oncologist. Some patients complete the intervention plan via Telehealth, which uses telecommunication technology to provide health services over a distance.
  Interventions: Other: Comprehensive Geriatric Assessment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration
- Arm II (standard of care) (Active Comparator): Patients follow a standard of care treatment plan at the discretion of the primary oncologist. Beginning 6 months from the start of chemotherapy, patients undergo the geriatric assessment as in Arm I. Some patients complete the standard of care treatment plan via Telehealth.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Follow geriatric assessment-driven treatment plan
  Arms: Arm I (geriatric assessment-driven treatment)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies a geriatric assessment intervention in predicting chemotherapy toxicity and vulnerabilities (or weakness) in older patients with cancer. Assessing patients' functional status, comorbidities, psychological state, social support, nutritional status, and cognitive function before treatment may help identify vulnerabilities, improve care, and decrease chemotherapy side effects in older patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify areas of vulnerability in older adults with cancer through the use of a geriatric assessment, and to identify the potential referrals to an interdisciplinary team based on geriatric assessment results.

II. To determine whether the geriatric assessment driven interventions will lead to decrease in grade 3-5 toxicity.

SECONDARY OBJECTIVES:

I. To determine whether the geriatric assessment driven interventions will lead to improvement in the following outcomes: unplanned hospitalization, average length of stay (ALOS), emergency visits, unplanned readmission rates, and advance directive completion.

II. To determine whether there is significantly better quality of life (QOL) and function in the geriatric assessment intervention group compared to the standard of care group from start of treatment to the follow-up timepoint.

III. To determine the feasibility of delivering geriatric assessment driven interventions in a community setting using telemedicine.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients follow an intervention plan created by the nurse practitioner (NP) using the results of the geriatric assessment. The NP discusses the results of the assessment and treatment recommendations with the patient. They also share the treatment plan, proposed referrals, and specific vulnerabilities with the primary care physician and community oncologist. Some patients complete the intervention plan via Telehealth, which uses telecommunication technology to provide health services over a distance.

ARM II: Patients follow a standard of care treatment plan at the discretion of the primary oncologist. Beginning 6 months from the start of chemotherapy, patients undergo the geriatric assessment as in Arm I. Some patients complete the standard of care treatment plan via Telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a solid tumor malignancy (any stage)
* Scheduled to start a new chemotherapy regimen (any line, combination cytotoxic chemotherapy with targeted agents are allowed)
* English, Spanish, and/or Chinese speaking
* Able to provide written informed consent

Exclusion Criteria:

* Not fluent in English, Spanish and/or Chinese (because not all questionnaires have been validated in other languages)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-08-04 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3-5 toxicity during chemotherapy | Up to 6 months
  Compared pre versus (vs) post-chemotherapy. Tested using general linear models with an alpha of 0.05.

SECONDARY OUTCOMES:
Rate of hospitalizations during chemotherapy | Up to 6 months
  Compared pre vs post-chemotherapy. General linear models will be considered for testing, but no alpha adjustments will be applied for multiple comparisons.
Change in functional status as measured by the Older American Resources and Services Instrumental Activities of Daily Living | Baseline to up to 6 months
  Compared pre vs post-chemotherapy. Explored using multivariate analyses. Results will be stratified by covariates such as patient age, poly- versus mono-chemotherapy, dose reduced or full dose therapy upfront, adjuvant versus metastatic disease, and number of prior chemotherapy regimens.
Change in quality of life as measured by Functional Assessment of Cancer Therapy - General | Baseline to up to 6 months
  Compared pre vs post-chemotherapy. Explored using multivariate analyses. Results will be stratified by covariates such as patient age, poly- versus mono-chemotherapy, dose reduced or full dose therapy upfront, adjuvant versus metastatic disease, and number of prior chemotherapy regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Daneng Li, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California

REFERENCES:
- [Derived] Li D, Sun CL, Kim H, Soto-Perez-de-Celis E, Chung V, Koczywas M, Fakih M, Chao J, Cabrera Chien L, Charles K, Hughes SFDS, Katheria V, Trent M, Roberts E, Jayani R, Moreno J, Kelly C, Sedrak MS, Dale W. Geriatric Assessment-Driven Intervention (GAIN) on Chemotherapy-Related Toxic Effects in Older Adults With Cancer: A Randomized Clinical Trial. JAMA Oncol. 2021 Nov 1;7(11):e214158. doi: 10.1001/jamaoncol.2021.4158. Epub 2021 Nov 18. PMID 34591080